CLINICAL TRIAL: NCT03515993
Title: Follow-up in Gynecological Cancer Survivors: An EORTC QLG-GCG Survivorship Study
Brief Title: Follow-up in Gynecological Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1514-QLG-GCG
Record Dates: First submitted 2018-03-30; First posted 2018-05-04 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Gynecologic Cancer
Keywords: long-term survival; gynecologic cancer; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional prospective study of follow-up in gynecologic cancer patients after primary treatment

DETAILED DESCRIPTION:
The objective of this study is to identify physical and psychosocial problems and needs after treatment for gynecological cancer.

1100 patients stratified by cancer sites and treatment - a minimum of 120 patients within each stratum - will be recruited.

Institutional data on follow-up policy, demographic and clinical data (related to treatment history and tumor characteristics) will be collected. Patients will complete a set of 76 Quality of Life questions, at one single time point.

Descriptive analyses will be conducted to characterize the collected data. Multivariate model building will be used to identify patterns of physical, psychological and social problems based on factors specific to the patient and to the disease. Logistic multinomial or continuous regression analysis will be used to investigate which socio-demographic, clinical variables, or institutional are associated significantly with compromised quality of life and sexual health outcomes. Exploratory factor analysis will be used to explore the factor structure of the various PROMs to identify issue clustering.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven gynecological cancer (cervical, endometrial, ovarian (including fallopian tube and peritoneal primary), vulva).
* FIGO stage I-IV before completion of primary therapy.
* Disease-free without any evidence of relapse: no symptoms or signs potentially indicating recurrent disease (assessed according to standard clinical parameters using physical and gynecological examination, blood tests, CA 125 (ovarian cancer), or radiological imaging techniques).
* At least 6 months but no more than 5 years since completion of primary treatment.
* Performance status 0, 1 or 2 (WHO scale).
* Age ≥ 18 years.
* Ability to understand and fill out questionnaires.
* Written informed consent according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Other cancer diagnosis in the past 5 years.
* Patients participating in interventional clinical studies with Quality of Life as primary endpoint.
* Any psychological (including pre-existing psychiatric disorders), familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Gynecologic cancer patients after primary treatment attending participating hospitals for routine follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | 15 months after first patient inclusion
  It will be evaluated using self-administered EORTC QLQ-C30 questionnaire
Health-related quality of life | 15 months after first patient inclusion
  It will be evaluated using self-administered questions on anxiety (from the EORTC quality of life item library)
Health-related quality of life | 15 months after first patient inclusion
  It will be evaluated using self-administered EORTC OUT-PATSAT-C7 questionnaire
Health-related quality of life | 15 months after first patient inclusion
  It will be evaluated using self-administered EORTC Sexual Health Questionnaire
Health-related quality of life | 15 months after first patient inclusion
  It will be evaluated using self-administered Distress Thermometer

CONTACTS AND LOCATIONS:
Locations (21):
- Medical University of Graz, Graz, Austria
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Chretien (CHC) - CHC MontLegia, Liège
  - ZNA Jan Palfijn, Merksem
- Germany (2):
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - HELIOS Kliniken - Helios Klinikum Wuppertal - Klin. Univ. Witten / Herdecke, Wuppertal
- Italy (3):
  - Ospedale San Gerardo, Monza
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- King Hussein Cancer Center, Amman, Jordan
- Netherlands (2):
  - Radboudumc - Radboud University Medical Center Nijmegen, Nijmegen
  - UMC-Academisch Ziekenhuis Utrecht, Utrecht
- Medical University Of Gdansk, Gdansk, Poland
- Spain (4):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
- United Kingdom (3):
  - East Kent Hospitals University NHS Foundation Trust - Queen Elizabeth The Queen Mother Hospita, Margate, Kent
  - Northampton General Hospital NHS Trust, Cliftonville, Northampton
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow